CLINICAL TRIAL: NCT01046617
Title: Lactobacillus Reuteri (DSM 17938) for the Treatment of Infantile Colic: a Randomized Double-blind Placebo Controlled Trial
Brief Title: Lactobacillus Reuteri for the Treatment of Infantile Colic:
Acronym: LRTIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Hania Szajewska, Department of Paediatrics, The Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 153/2009
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Infantile Colic; Crying
Keywords: infantile colic; Lactobacillus reuteri; duration of crying
MeSH Terms: conditions — Colic; Crying

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri (DSM 17938) — 5 drops once daily (10(8) CFU) for 21 days

SUMMARY:
Infantile colic is characterized by excessive crying (defined as crying that last at least 3 hours a day, for 3 days a week, for at least 3 weeks) in an otherwise healthy infant. The crying typically starts in the first few weeks of life and ends by 4-5 months of age. The condition is usually self-limited, with no long-term adverse effects; however, it may be very distressing to parents, hence, any safe and effective treatment would be desirable. Recently, it has been suggested that probiotics may offer some benefit.This is based on the results of one open randomized controlled trial. In this trial, 83 breast-fed infants with colic defined as >3 hours of crying on >3 days/week were randomly allocated to receive Lactobacillus reuteri DSM 17938 (108 colony-forming units, once daily 30 minutes after feeding) or simethicone (60 mg/day as 15 drops twice a day after feeding) for 28 days. Mothers followed a cow's milk free diet. By day 28 after randomization, mothers of infants in the probiotic group were significantly more likely than mothers of infants in the simethicone group to report a reduction from baseline in average crying time to less than 3 hours per day (95% vs. 7%). In addition, median crying times were significantly shorter in the probiotic group than in the simethicone group. No adverse effects of L. reuteri were reported.

Although the mechanism of action of L. reuteri for treating infantile colic has not been elucidated yet, the findings are very promising. However, there are some methodological limitations to the study, including no allocation concealment, no blinding, and no intention-to-treat analysis; these may result in selection, performance, and/or attrition biases and, eventually, invalidate the results. Another limitation of the study is the lack of a true placebo group. Given these consideration a new study is proposed that is aiming to overcome these limitations.

DETAILED DESCRIPTION:
Eligible infants will be randomly assigned to receive either L. reuteri 108 CFU per day or placebo. Both the active treatment and placebo will be taken orally, 1 times daily, for 21 days.

All infants are eligible for screening. If a patient appears to meet the criteria for enrollment and express interest in the study, cow's milk elimination diet will be prescribed for 1 week to a breastfeeding mother (and to an infant, in case of formula fed infants). Care givers will be asked to record for 1 week symptoms of colic. Children fulfilling inclusion criteria will be asked to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Full-term infants age <5 months
* Infantile colic (>3 hours of crying on >3 days in the week) within 7 days prior to enrollment
* Exclusive or predominant (>50%) breastfeeding
* Informed consent

Exclusion Criteria:

* Acute or chronic illness
* Gastrointestinal disorders
* Use of any antibiotics and/or probiotic pharmaceutical products within 7 days prior to the study.

Ages: 1 Month to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Duration of crying (minutes per day) | 21 days
Reduction on the daily average crying time >50% during the study | 21 days

SECONDARY OUTCOMES:
Reduction of the daily average crying time, from baseline to the end of the treatment period, to <3 hours/day | 21 days
Persistence of infantile colic after the intervention | 21 days
Parental perception of severity | 21 days
Parental or family quality of life | 21 days
Growth parameters | 21 days
Adverse effects (e.g. vomiting, constipation, etc.) | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical University of Warsaw, Outpatient Clinic, Warsaw, Poland

REFERENCES:
- [Derived] Szajewska H, Gyrczuk E, Horvath A. Lactobacillus reuteri DSM 17938 for the management of infantile colic in breastfed infants: a randomized, double-blind, placebo-controlled trial. J Pediatr. 2013 Feb;162(2):257-62. doi: 10.1016/j.jpeds.2012.08.004. Epub 2012 Sep 14. PMID 22981952